CLINICAL TRIAL: NCT00351910
Title: A Multi-Centre, Double-Blind, Randomised, Parallel-Group, Placebo-Controlled Phase III Study of the Efficacy and Safety of Quetiapine Fumarate Sustained Release (Seroquel SRTM) in Combination With an Antidepressant in the Treatment of Patients With Major Depressive Disorder With Inadequate Response to an Antidepressant Treatment
Brief Title: Efficacy of Seroquel SR in Combination With an Antidepressant in Treatment of Major Depressive Disorder
Acronym: ONYX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1448C00007; ONYX; EUDRACT No: 2005-0055053-22
Record Dates: First submitted 2006-07-12; First posted 2006-07-13 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Quetiapine Fumarate; Amitriptyline; Bupropion; Citalopram; Duloxetine Hydrochloride; Escitalopram; Fluoxetine; Paroxetine; Sertraline; Venlafaxine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Quetiapine
Drug: Amitriptyline
Drug: Bupropion
Drug: Citalopram
Drug: Duloxetine
Drug: Escitalopram
Drug: Fluoxetine
Drug: Paroxetine
Drug: Sertraline
Drug: Venlafaxine

SUMMARY:
To evaluate the efficacy of quetiapine fumarate sustained release (Seroquel SR™) in combination with an antidepressant versus an antidepressant alone in patients with Major Depressive Disorder.

PLEASE NOTE: Seroquel SR and Seroquel XR refer to the same formulation. The SR designation was changed to XR after consultation with FDA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 65 years
* A documented diagnosis of major depressive disorder

Exclusion Criteria:

* Patients with a DSM IV Axis I disorder other than MDD within 6 months of enrolment
* Patients with a diagnosis of DSM IV Axis II disorder which has a major impact on the patient's current psychiatric status
* Patients whose current episode of depression exceeds 12 months or is less than 4 weeks prior to enrolment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Actual)
Dates: Start 2006-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the efficacy of quetiapine fumarate sustained release
(Seroquel SR™) in combination with an antidepressant versus an antidepressant alone in patients with Major Depressive Disorder.

SECONDARY OUTCOMES:
If quetiapine SR in combination with an antidepressant improves health-related quality of life of patients with MDD, compared to an antidepressant alone.

CONTACTS AND LOCATIONS:
Overall Officials: Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (72):
- Australia (7):
  - Research Site, Everton Park, Queensland
  - Research Site, Southport, Queensland
  - Research Site, Frankston, Victoria
  - Research Site, Malvern, Victoria
  - Research Site, Prahran, Victoria
  - Research Site, Richmond, Victoria
  - Research Site, Brisbane
- Belgium (7):
  - Research Site, Assebroek
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Kortrijk
  - Research Site, Liège
  - Research Site, Mechelen
  - Research Site, Tielt
- Canada (7):
  - Research Site, Edmonton, Alberta
  - Research Site, Moncton, New Brunswick
  - Research Site, Mount Pearl, Newfoundland and Labrador
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Toronto, Ontario
  - Research Site, Pointe-Claire, Quebec
- Czechia (7):
  - Research Site, Brno
  - Research Site, Havířov
  - Research Site, Havlíčkův Brod
  - Research Site, Nové Město nad Metují
  - Research Site, Olomouc
  - Research Site, Ostrava
  - Research Site, Prague
- Finland (4):
  - Research Site, Helsinki
  - Research Site, Jarvenpaa
  - Research Site, Salo
  - Research Site, Turku
- France (10):
  - Research Site, Angoulême
  - Research Site, Arcachon
  - Research Site, Caen
  - Research Site, Château-Gontier
  - Research Site, Élancourt
  - Research Site, Le Pecq
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Toulouse
- Germany (4):
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Münster
- Norway (7):
  - Research Site, Bergen
  - Research Site, Flekkefjord
  - Research Site, Fyllingsdalen
  - Research Site, Hamar
  - Research Site, Lysaker
  - Research Site, Oslo
  - Research Site, Skien
- Poland (6):
  - Research Site, Gdansk
  - Research Site, Lodz
  - Research Site, Nowy Targ
  - Research Site, Szczecin
  - Research Site, Torun
  - Research Site, Warsaw
- Romania (2):
  - Research Site, Bucharest
  - Research Site, Piteşti
- South Africa (3):
  - Research Site, Pretoria, Gauteng
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Cape Town, Western Cape
- Sweden (8):
  - Research Site, Falköping
  - Research Site, Gothenburg
  - Research Site, Halmstad
  - Research Site, Malmo
  - Research Site, Stockholm
  - Research Site, Sundsvall
  - Research Site, Trollhättan
  - Research Site, Uppsala

REFERENCES:
- [Derived] McIntyre RS, Gorwood P, Thase ME, Liss C, Desai D, Chen J, Bauer M. Early Symptom Improvement as a Predictor of Response to Extended Release Quetiapine in Major Depressive Disorder. J Clin Psychopharmacol. 2015 Dec;35(6):706-10. doi: 10.1097/JCP.0000000000000416. PMID 26474010
- [Derived] Weisler R, Montgomery SA, Earley WR, Szamosi J, Eriksson H. Extended release quetiapine fumarate in patients with major depressive disorder: suicidality data from acute and maintenance studies. J Clin Psychiatry. 2014 May;75(5):520-7. doi: 10.4088/JCP.13m08624. PMID 24816198
- [Derived] Weisler R, McIntyre RS, Bauer M. Extended-release quetiapine fumarate in the treatment of patients with major depressive disorder: adjunct therapy. Expert Rev Neurother. 2013 Nov;13(11):1183-200. doi: 10.1586/14737175.2013.846519. PMID 24175721
- [Derived] Bauer M, Demyttenaere K, El-Khalili N, Thase ME, Papakostas GI, Szamosi J, Earley WR, Eriksson H. Pooled analysis of adjunct extended-release quetiapine fumarate in patients with major depressive disorder according to ongoing SSRI or SNRI treatment. Int Clin Psychopharmacol. 2014 Jan;29(1):16-25. doi: 10.1097/YIC.0000000000000011. PMID 24108148
- [Derived] Clayton AH, Locklear JC, Svedsater H, McIntyre RS. Sexual functioning in patients with major depressive disorder in randomized placebo-controlled studies of extended release quetiapine fumarate. CNS Spectr. 2014 Apr;19(2):182-96. doi: 10.1017/S1092852913000631. Epub 2013 Sep 25. PMID 24067192
- [Derived] Bauer M, McIntyre RS, Szamosi J, Eriksson H. Evaluation of adjunct extended-release quetiapine fumarate on sleep disturbance and quality in patients with major depressive disorder and an inadequate response to on-going antidepressant therapy. Int J Neuropsychopharmacol. 2013 Sep;16(8):1755-65. doi: 10.1017/S146114571300031X. Epub 2013 May 14. PMID 23672772
- [Derived] Vieta E, Bauer M, Montgomery S, McIntyre RS, Szamosi J, Earley WR, Eriksson H. Pooled analysis of sustained response rates for extended release quetiapine fumarate as monotherapy or adjunct to antidepressant therapy in patients with major depressive disorder. J Affect Disord. 2013 Sep 5;150(2):639-43. doi: 10.1016/j.jad.2013.01.052. Epub 2013 Mar 14. PMID 23497790
- [Derived] Bauer M, Pretorius HW, Constant EL, Earley WR, Szamosi J, Brecher M. Extended-release quetiapine as adjunct to an antidepressant in patients with major depressive disorder: results of a randomized, placebo-controlled, double-blind study. J Clin Psychiatry. 2009 Apr;70(4):540-9. doi: 10.4088/jcp.08m04629. Epub 2009 Apr 7. PMID 19358791